CLINICAL TRIAL: NCT02552316
Title: The Cutaneous Microbiota of Psoriasis: Lesional Variation and a Phase IV, Interventional Study of Its Response to Phototherapy
Brief Title: Psoriasis Microbiome and Phototherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 821876
Record Dates: First submitted 2015-09-09; First posted 2015-09-17 (Estimated); Results first posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Psoriasis
Keywords: microbiome; bacteria; NB-UVB Phototherapy; light therapy
MeSH Terms: conditions — Psoriasis | interventions — Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NB-UVB Phototherapy (Other): NB-UVB phototherapy is a therapy which uses ultraviolet B (UVB) light directed at the skin. This type of light therapy is given through the use of phototherapy booths which contain fluorescent tubes that emit UVB light. Booths used for phototherapy look similar to commercial tanning booths. NB-UVB phototherapy affects psoriasis by causing changes to the cells of the skin and producing a local effect by reducing the number of certain types of skin cells which have an impact on psoriasis formation.
  Interventions: Device: NB-UVB Phototherapy

INTERVENTIONS:
Device: NB-UVB Phototherapy
  Other Names: Phototherapy; Light therapy

SUMMARY:
The ASPIRE study is a clinical trial designed to examine the microbes (e.g., bacteria) within psoriasis skin lesions compared with normal skin. The investigators will also examine the effect of NB-UVB (narrow-band ultraviolet B) phototherapy (i.e., light therapy) on skin microbes.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 years of age and older.
2. Clinical diagnosis of psoriasis for at least 6 months as determined by subject interview of his/her medical history and confirmation of diagnosis through physical examination by Investigator.
3. Stable plaque psoriasis for at least 2 months before Screening and at Baseline (Week 1) as determined by subject interview of his/her medical history.
4. Subject is a candidate for phototherapy.
5. Subject has at least one psoriatic plaque measuring at least 6cm x 2cm located on either the arms or the legs (excluding intertriginous areas such as the axilla and inguinal folds)
6. Able and willing to give written informed consent and to comply with requirements of this study protocol.

Exclusion Criteria:

1. Subject has photosensitizing condition or other contraindication to phototherapy
2. Diagnosis of erythrodermic psoriasis, generalized or localized pustular psoriasis, medication-induced or medication-exacerbated psoriasis, or new onset guttate psoriasis.
3. Cannot discontinue or avoid topical therapies for psoriasis for at least 14 days prior to the Baseline (Week 1) visit and during the study other than on face, underarms, or groin.
4. Cannot discontinue or avoid UVB phototherapy or Excimer laser for at least 14 days prior to the Baseline (Week 1) visit.
5. Subject is receiving therapy for psoriasis that requires a wash out period of more than 14 days (e.g., psoralen-UVA phototherapy, oral systemic therapy, biologic therapy, or other investigational therapy).
6. Other active inflammatory dermatologic conditions (e.g., eczema) or presence of pustular or erythrodermic psoriasis.
7. Any history of acute or chronic bacterial, fungal, or viral infection (including HIV, hepatitis, tuberculosis, or other severe or recurrent infections) within 30 days of baseline sample collection.
8. Subject has used systemic (oral or parenteral) antibiotic, antimycotic, or antiviral within 3 months or topical antibiotic, antimycotic, or antiviral within 14 days of baseline sample collection or requires use of any topical or systemic antibiotic, antimycotic, or antiviral during the study.
9. Consumption of large doses of commercial probiotics (greater than or equal to 108 cfu or organisms per day) including tablets, capsules, lozenges, chewing gum or powders in which probiotic is a primary component. Ordinary dietary components such as fermented beverages/milks, yogurts, and foods do not apply.
10. Presence of comorbid medical condition (e.g., HIV, malignancy within past 5 years other than successfully treated basal cell carcinoma, non-metastatic cutaneous squamous cell carcinoma or cervical carcinoma in-situ) that significantly alters the immune system or results in immunosuppression.
11. Subject is taking (within up to 180 days of baseline sample collection) or requires topical or systemic therapy during the study that significantly alters the immune system or results in immunosuppression (e.g., chemotherapy, oral or injectable corticosteroid). Inhaled corticosteroids for stable medical conditions are allowed.
12. Unstable dietary history as defined by major changes in diet within 30 days of baseline or during study, where the subject has or plans to eliminate or significantly increase major food group in the diet.
13. Recent history of substance abuse or psychiatric illness that could preclude compliance with the protocol.
14. History of any substance abuse within 365 days of screening visit.
15. Female subject who is pregnant or breast-feeding or considering becoming pregnant during the study.
16. Major surgery of the gastrointestinal tract, with the exception of cholecystectomy and appendectomy, in the past 5 years. Any major bowel resection at any time.
17. History of active uncontrolled gastrointestinal disorders or diseases including:

    * Inflammatory bowel disease including ulcerative colitis, Crohn's disease, or indeterminate colitis;
    * Irritable bowel syndrome;
    * Persistent, infectious gastroenteritis, colitis, or gastritis, persistent or chronic diarrhea or unknown etiology, Clostridium difficile infection (recurrent) or Helicobacter pylori infection (untreated).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2020-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Junko Takeshita, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- NB-UVB Phototherapy: Narrow band-UVB (NB-UVB) phototherapy is a therapy which uses ultraviolet B (UVB) light directed at the skin. This type of light therapy is given through the use of phototherapy booths which contain fluorescent tubes that emit UVB light. Booths used for phototherapy look similar to commercial tanning booths. NB-UVB phototherapy affects psoriasis by causing changes to the cells of the skin and producing a local effect by reducing the number of certain types of skin cells which have an impact on psoriasis formation.
  In the study, NB-UVB phototherapy administered 3 times per week for 8 weeks.
Period: Overall Study
Arm/Group | NB-UVB Phototherapy
Started | 34
Completed | 32
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Withdrawal due to non-compliance | 1

BASELINE CHARACTERISTICS:
Groups:
- NB-UVB Phototherapy: NB-UVB phototherapy is a therapy which uses ultraviolet B (UVB) light directed at the skin. This type of light therapy is given through the use of phototherapy booths which contain fluorescent tubes that emit UVB light. Booths used for phototherapy look similar to commercial tanning booths. NB-UVB phototherapy affects psoriasis by causing changes to the cells of the skin and producing a local effect by reducing the number of certain types of skin cells which have an impact on psoriasis formation.
  NB-UVB Phototherapy
Arm/Group | NB-UVB Phototherapy
Number analyzed (Participants) | 34
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 45.5 [30 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 22
  More than one race | 0
  Unknown or Not Reported | 2
Body Mass Index [Median (Inter-Quartile Range); unit: Kg/m^2] | 29.60 [23.88 to 34.66]
Fitzpatrick skin type [Count of Participants; unit: Participants] — Fitzpatrick skin type describes a method of classifying skin by its reaction to sunlight. This system classifies skin types from I through V whereby a lower Fitzpatrick skin type classification indicates skin that burns more easily than it tans, while a higher Fitzpatrick skin type indicates the opposite. The skin type classification criteria are detailed below.
  Type I: Always burns, never tans Type II: Burns easily, tans poorly Type III: Tans after initial burn Type IV: Rarely burns and tans darkly easily Type V: Never burns, always tans very darkly
  Participants
    Type I | 1
    Type II | 18
    Type III | 6
    Type IV | 4
    Type V | 5
Age of psoriasis onset [Count of Participants; unit: Participants]
  < 20 years | 16
  20 - 39 years | 10
  ≥40 years | 8
Duration of psoriasis (year) [Median (Inter-Quartile Range); unit: years] | 11.5 [7 to 22]
Psoriasis Area and Severity Index (PASI) score [Median (Inter-Quartile Range); unit: units on a scale] — The Psoriasis Area Severity Index (PASI) is an instrument that measures the severity and extent of psoriasis. The score is based on a combination of psoriasis appearance (erythema, induration and desquamation) and percentage of body surface area. The scale ranges from 0 (no disease) to 72 (maximal disease severity), whereby higher PASI scores indicate higher severity of psoriasis.
  units on a scale | 9.55 [7.6 to 14.3]
Physician Global Assessment (PGA) [Median (Inter-Quartile Range); unit: units on a scale] — This PGA scale is an assessment of severity whereby physician's rating of erythema, induration and scaling is assessed, individually, on a five-point scale (from 0 = no symptom to 4 = severe). The total score is the mean of the three item scores, each having an equal weighting, with the total scores ranging between 0 (clear skin) and 4 (severe disease) and higher score indicating more severe psoriasis.
  units on a scale
    Overall | 3 [2.7 to 3.3]
    Lesion | 3 [3 to 3.7]
Body Surface Area (BSA) [Median (Inter-Quartile Range); unit: percentage (%)] | 7.55 [5 to 10.25]
Psoriatic arthritis diagnosis [Count of Participants; unit: Participants]
  No | 33
  Yes | 1
Plaque location [Count of Participants; unit: Participants]
  Arm | 8
  Leg | 26

OUTCOME MEASURES:

1. Primary Outcome: Cutaneous Microbiota Shannon's Alpha Diversity at Baseline
Description: Variation in the microbial diversity of skin affected and unaffected by psoriasis was characterized at baseline.
  The Alpha Diversity Index is a quantitative measure that reflects the diversity of bacterial species in a sample. The greater the index value, the more diverse the skin microbiota. The diversity of the microbiota present in the given sample was measured using the Shannon Diversity Index, whereby each "arm title" is describing the difference in the measure of diversity between the comparison groups.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: Shannon's index
Groups:
- Group 1a- Plaque Center vs Plaque Edge: The diversity of microbiota present in a given sample measured using the Shannon Diversity Index at baseline prior to initiation of phototherapy.
  Difference in the measure of Shannon diversity index between plaque center vs plaque edge.
- Group 1b- Plaque Center vs Ipsilateral Perilesional Unaffected: The diversity of microbiota present in a given sample measured using the Shannon Diversity Index at baseline prior to initiation of phototherapy.
  Difference in the measure of Shannon diversity index between plaque center vs ipsilateral perilesional unaffected skin
- Group 1c- Plaque Center vs Ipsilateral Distant Unaffected Skin: The diversity of microbiota present in a given sample measured using the Shannon Diversity Index at baseline prior to initiation of phototherapy.
  Difference in the measure of Shannon diversity index between plaque center vs ipsilateral distant unaffected skin.
- Group 1d- Ipsilateral Unaffected Skin: Perilesional vs Distant: The diversity of microbiota present in a given sample measured using the Shannon Diversity Index at baseline prior to initiation of phototherapy.
  Difference in the measure of Shannon diversity index between perilesional ipsilateral unaffected skin vs distant ipsilateral unaffected skin.
- Group 1e- Plaque Center vs Contralateral Unaffected Skin: The diversity of microbiota present in a given sample measured using the Shannon Diversity Index at baseline prior to initiation of phototherapy.
  Difference in the measure of Shannon diversity index between plaque center vs contralateral unaffected skin.
Arm/Group | Group 1a- Plaque Center vs Plaque Edge | Group 1b- Plaque Center vs Ipsilateral Perilesional Unaffected | Group 1c- Plaque Center vs Ipsilateral Distant Unaffected Skin | Group 1d- Ipsilateral Unaffected Skin: Perilesional vs Distant | Group 1e- Plaque Center vs Contralateral Unaffected Skin
Number analyzed (Participants) | 15 | 24 | 26 | 29 | 10
Shannon's index | -0.05 (0.06) | 0.06 (0.10) | -0.06 (0.09) | 0.12 (0.08) | 0.26 (0.12)

2. Primary Outcome: Change in Cutaneous Microbiota Shannon's Alpha Diversity at Baseline vs Week 8
Description: Variation in the microbial diversity of skin affected and unaffected by psoriasis was characterized at baseline. Changes in microbial diversity was assessed between baseline and week 8.
  The Alpha Diversity Index is a quantitative measure that reflects the diversity of bacterial species in a sample. The greater the index value, the more diverse the skin microbiota. The diversity of the microbiota present in the given sample was measured using the Shannon Diversity Index, whereby each "arm title" is describing the difference in the measure of diversity between the comparison groups.
Time Frame: Week 8
Measure: Mean (Standard Error); unit: Shannon's index
Groups:
- Group 2a- Plaque Center: The diversity of microbiota present in a given sample measured using the Shannon Diversity Index at baseline prior to initiation of phototherapy and week 8 after initiation of phototherapy.
  Difference in the measure of Shannon diversity index between plaque center at baseline vs week 8.
- Group 2b- Ipsilateral Distant Unaffected Skin: The diversity of microbiota present in a given sample measured using the Shannon Diversity Index at baseline prior to initiation of phototherapy and week 8 after initiation of phototherapy.
  Difference in the measure of Shannon diversity index between ipsilateral distant unaffected skin at baseline vs week 8.
- Group 2c- Contralateral Unaffected Skin: The diversity of microbiota present in a given sample measured using the Shannon Diversity Index at baseline prior to initiation of phototherapy and week 8 after initiation of phototherapy.
  Difference in the measure of Shannon diversity index between contralateral unaffected skin at baseline vs week 8.
- Group 2d- Unaffected Back Skin: The diversity of microbiota present in a given sample measured using the Shannon Diversity Index at baseline prior to initiation of phototherapy and week 8 after initiation of phototherapy.
  Difference in the measure of Shannon diversity index between unaffected back skin at baseline vs week 8.
Arm/Group | Group 2a- Plaque Center | Group 2b- Ipsilateral Distant Unaffected Skin | Group 2c- Contralateral Unaffected Skin | Group 2d- Unaffected Back Skin
Number analyzed (Participants) | 26 | 25 | 12 | 30
Shannon's index | -0.08 (0.12) | -0.12 (0.11) | 0.03 (0.16) | -0.07 (0.13)

3. Primary Outcome: Change in Cutaneous Microbiota Shannon's Alpha Diversity at Baseline vs Week 9.
Description: Variation in the microbial diversity of skin affected and unaffected by psoriasis was characterized at baseline. Changes in microbial diversity was assessed between baseline and week 9.
  The Alpha Diversity Index is a quantitative measure that reflects the diversity of bacterial species in a sample. The greater the index value, the more diverse the skin microbiota. The diversity of the microbiota present in the given sample was measured using the Shannon Diversity Index, whereby each "arm title" is describing the difference in the measure of diversity between the comparison groups.
Time Frame: Week 9
Measure: Mean (Standard Error); unit: Shannon's index
Groups:
- Group 3a- Plaque Center: The diversity of microbiota present in a given sample measured using the Shannon Diversity Index at baseline prior to initiation of phototherapy and week 9 after initiation of phototherapy.
  Difference in the measure of Shannon diversity index between plaque center at baseline vs week 9.
- Group 3b- Ipsilateral Distant Unaffected Skin: The diversity of microbiota present in a given sample measured using the Shannon Diversity Index at baseline prior to initiation of phototherapy and week 9 after initiation of phototherapy.
  Difference in the measure of Shannon diversity index between ipsilateral distant unaffected skin at baseline vs week 9.
- Group 3c- Contralateral Unaffected Skin: The diversity of microbiota present in a given sample measured using the Shannon Diversity Index at baseline prior to initiation of phototherapy and week 9 after initiation of phototherapy.
  Difference in the measure of Shannon diversity index between contralateral unaffected skin at baseline vs week 9.
- Group 3d- Unaffected Back Skin: The diversity of microbiota present in a given sample measured using the Shannon Diversity Index at baseline prior to initiation of phototherapy and week 9 after initiation of phototherapy.
  Difference in the measure of Shannon diversity index between unaffected back skin at baseline vs week 9.
Arm/Group | Group 3a- Plaque Center | Group 3b- Ipsilateral Distant Unaffected Skin | Group 3c- Contralateral Unaffected Skin | Group 3d- Unaffected Back Skin
Number analyzed (Participants) | 26 | 25 | 11 | 31
Shannon's index | -0.03 (0.11) | -0.13 (0.16) | -0.01 (0.16) | 0.19 (0.11)

4. Primary Outcome: Cutaneous Microbiota Jaccard's Beta Diversity at Baseline
Description: Variation in the microbial diversity of skin affected and unaffected by psoriasis was characterized at baseline.
  The Beta Diversity Index is a quantitative measure that reflects the diversity of bacterial species between two different regions. The greater the index, the more diverse the microbiota between the two regions.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: Jaccard index
Groups:
- Group 1: The diversity of microbiota present in a given sample measured using the Jaccard's Diversity Index at baseline prior to initiation of phototherapy.
  Comparison of differences in mean between plaque edge vs plaque center and ipsilateral perilesional unaffected skin vs plaque center at baseline.
- Group 2: The diversity of microbiota present in a given sample measured using the Jaccard's Diversity Index at baseline prior to initiation of phototherapy.
  Comparison of differences in mean between plaque edge vs plaque center and ipsilateral distant unaffected skin vs plaque center at baseline.
- Group 3: The diversity of microbiota present in a given sample measured using the Jaccard's Diversity Index at baseline prior to initiation of phototherapy.
  Comparison of differences in mean between plaque edge vs plaque center and contralateral unaffected skin vs plaque center at baseline.
- Group 4: The diversity of microbiota present in a given sample measured using the Jaccard's Diversity Index at baseline prior to initiation of phototherapy.
  Comparison of differences in mean between Ipsilateral perilesional unaffected skin vs plaque center and ipsilateral distant unaffected skin vs plaque center at baseline.
- Group 5: The diversity of microbiota present in a given sample measured using the Jaccard's Diversity Index at baseline prior to initiation of phototherapy.
  Comparison of differences in mean between Ipsilateral perilesional unaffected skin vs plaque center and contralateral unaffected skin vs plaque center at baseline.
- Group 6: The diversity of microbiota present in a given sample measured using the Jaccard's Diversity Index at baseline prior to initiation of phototherapy.
  Comparison of differences in mean between Ipsilateral distant unaffected skin vs plaque center and contralateral unaffected skin vs plaque center at baseline.
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Number analyzed (Participants) | 24 | 27 | 20 | 27 | 26 | 27
Jaccard index | 0.003 (0.015) | 0.012 (0.014) | 0.021 (0.015) | 0.009 (0.010) | 0.018 (0.011) | 0.009 (0.010)

5. Primary Outcome: Change in Cutaneous Microbiota Jaccard's Beta Diversity at Baseline vs Week 8
Description: Variation in the microbial diversity of skin affected and unaffected by psoriasis was characterized at baseline. Changes in microbial diversity was assessed between baseline and week 8.
  The Beta Diversity Index is a quantitative measure that reflects the diversity of bacterial species between two different regions. The greater the index, the more diverse the microbiota between the two regions.
Time Frame: Week 8
Measure: Mean (Standard Error); unit: Jaccard's index
Groups:
- Plaque Edge vs Center: The diversity of microbiota present in a given sample measured using the Jaccard's Diversity Index at baseline prior to initiation of phototherapy and week 8 after initiation of phototherapy.
  Comparison of differences in mean between plaque edge vs plaque center at baseline vs plaque edge vs plaque center at week 8.
- Ipsilateral Perilesional Unaffected Skin vs Plaque Center: The diversity of microbiota present in a given sample measured using the Jaccard's Diversity Index at baseline prior to initiation of phototherapy and week 8 after initiation of phototherapy.
  Comparison of differences in mean between Ipsilateral perilesional unaffected skin vs plaque center at baseline vs Ipsilateral perilesional unaffected skin vs plaque center at week 8.
- Ipsilateral Distant Unaffected Skin vs Plaque Center: The diversity of microbiota present in a given sample measured using the Jaccard's Diversity Index at baseline prior to initiation of phototherapy and week 8 after initiation of phototherapy.
  Comparison of differences in mean between Ipsilateral distant unaffected skin vs plaque center at baseline vs Ipsilateral distant unaffected skin vs plaque center at week 8.
- Contralateral Unaffected Skin vs Plaque Center: The diversity of microbiota present in a given sample measured using the Jaccard's Diversity Index at baseline prior to initiation of phototherapy and week 8 after initiation of phototherapy.
  Comparison of differences in mean between contralateral unaffected skin vs plaque center at baseline vs contralateral unaffected skin vs plaque center at week 8.
- Unaffected Back vs Plaque Center: The diversity of microbiota present in a given sample measured using the Jaccard's Diversity Index at baseline prior to initiation of phototherapy and week 8 after initiation of phototherapy.
  Comparison of differences in mean between unaffected back vs plaque center at baseline vs unaffected back vs plaque center at week 8.
Arm/Group | Plaque Edge vs Center | Ipsilateral Perilesional Unaffected Skin vs Plaque Center | Ipsilateral Distant Unaffected Skin vs Plaque Center | Contralateral Unaffected Skin vs Plaque Center | Unaffected Back vs Plaque Center
Number analyzed (Participants) | 15 | 29 | 29 | 15 | 32
Jaccard's index | -0.021 (0.020) | -0.002 (0.016) | 0.008 (0.009) | 0.013 (0.011) | 0.008 (0.010)

6. Primary Outcome: Change in Cutaneous Microbiota Jaccard's Beta Diversity at Baseline vs Week 9
Description: Variation in the microbial diversity of skin affected and unaffected by psoriasis was characterized at baseline. Changes in microbial diversity was assessed between baseline and week 9.
  The Beta Diversity Index is a quantitative measure that reflects the diversity of bacterial species between two different regions. The greater the index, the more diverse the microbiota between the two regions.
Time Frame: Week 9
Measure: Mean (Standard Error); unit: Jaccard's index
Groups:
- Plaque Edge vs Center: The diversity of microbiota present in a given sample measured using the Jaccard's Diversity Index at baseline prior to initiation of phototherapy and week 9 after initiation of phototherapy.
  Comparison of differences in mean between plaque edge vs plaque center at baseline vs plaque edge vs plaque center at week 9.
- Ipsilateral Perilesional Unaffected Skin vs Plaque Center: The diversity of microbiota present in a given sample measured using the Jaccard's Diversity Index at baseline prior to initiation of phototherapy and week 9 after initiation of phototherapy.
  Comparison of differences in mean between Ipsilateral perilesional unaffected skin vs plaque center at baseline vs Ipsilateral perilesional unaffected skin vs plaque center at week 9.
- Ipsilateral Distant Unaffected Skin vs Plaque Center: The diversity of microbiota present in a given sample measured using the Jaccard's Diversity Index at baseline prior to initiation of phototherapy and week 9 after initiation of phototherapy.
  Comparison of differences in mean between Ipsilateral distant unaffected skin vs plaque center at baseline vs Ipsilateral distant unaffected skin vs plaque center at week 9.
- Contralateral Unaffected Skin vs Plaque Center: The diversity of microbiota present in a given sample measured using the Jaccard's Diversity Index at baseline prior to initiation of phototherapy and week 9 after initiation of phototherapy.
  Comparison of differences in mean between contralateral unaffected skin vs plaque center at baseline vs contralateral unaffected skin vs plaque center at week 9.
- Unaffected Back vs Plaque Center: The diversity of microbiota present in a given sample measured using the Jaccard's Diversity Index at baseline prior to initiation of phototherapy and week 9 after initiation of phototherapy.
  Comparison of differences in mean between unaffected back vs plaque center at baseline vs unaffected back vs plaque center at week 9.
Arm/Group | Plaque Edge vs Center | Ipsilateral Perilesional Unaffected Skin vs Plaque Center | Ipsilateral Distant Unaffected Skin vs Plaque Center | Contralateral Unaffected Skin vs Plaque Center | Unaffected Back vs Plaque Center
Number analyzed (Participants) | 15 | 28 | 29 | 15 | 32
Jaccard's index | -0.016 (0.019) | -0.001 (0.010) | -0.007 (0.009) | -0.004 (0.011) | 0.0002 (0.011)

7. Primary Outcome: Cutaneous Bacterial Load at Baseline
Description: Bacterial count per sample at baseline prior to initiation of phototherapy.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: Log10 [bacterial count/sample]
Groups:
- Plaque Edge vs Center: Bacterial load in a given sample using log10 (bacterial count/ sample) units at baseline prior to initiation of phototherapy.
  Comparison between plaque edge vs plaque center at baseline.
- Ipsilateral Perilesional Unaffected Skin vs Plaque Center: Bacterial load in a given sample using log10 (bacterial count/ sample) units at baseline prior to initiation of phototherapy.
  Comparison between Ipsilateral perilesional unaffected skin vs plaque center at baseline.
- Ipsilateral Distant Unaffected Skin vs Plaque Center: Bacterial load in a given sample using log10 (bacterial count/ sample) units at baseline prior to initiation of phototherapy.
  Comparison between Ipsilateral distant unaffected skin vs plaque center at baseline.
- Contralateral Unaffected Skin vs Plaque Center: Bacterial load in a given sample using log10 (bacterial count/ sample) units at baseline prior to initiation of phototherapy.
  Comparison between contralateral unaffected skin vs plaque center at baseline.
Arm/Group | Plaque Edge vs Center | Ipsilateral Perilesional Unaffected Skin vs Plaque Center | Ipsilateral Distant Unaffected Skin vs Plaque Center | Contralateral Unaffected Skin vs Plaque Center
Number analyzed (Participants) | 34 | 34 | 34 | 34
Log10 [bacterial count/sample] | 0.21 (0.24) | 0.60 (0.18) | 0.71 (0.17) | 0.57 (0.21)

8. Primary Outcome: Change in Cutaneous Bacterial Load Between Baseline and Week 8.
Description: Bacterial count per sample at baseline prior to initiation of phototherapy vs at week 8 after initiation of phototherapy.
Time Frame: Week 8
Measure: Mean (Standard Error); unit: Log10 [bacterial count/sample]
Groups:
- Plaque Center: Change in bacterial load in a given sample using log10 (bacterial count/ sample) units at baseline prior to initiation of phototherapy and at week 8 after the initiation of phototherapy.
  Comparison between plaque center at baseline vs plaque center at week 8.
- Plaque Edge: Change in bacterial load in a given sample using log10 (bacterial count/ sample) units at baseline prior to initiation of phototherapy and at week 8 after the initiation of phototherapy.
  Comparison between plaque edge at baseline vs plaque edge at week 8.
- Ipsilateral Perilesional Unaffected Skin: Change in bacterial load in a given sample using log10 (bacterial count/ sample) units at baseline prior to initiation of phototherapy and at week 8 after the initiation of phototherapy.
  Comparison between ipsilateral perilesional unaffected skin at baseline vs ipsilateral perilesional unaffected skin at week 8.
- Ipsilateral Distant Unaffected Skin: Change in bacterial load in a given sample using log10 (bacterial count/ sample) units at baseline prior to initiation of phototherapy and at week 8 after the initiation of phototherapy.
  Comparison between ipsilateral distant unaffected skin at baseline vs ipsilateral distant unaffected skin at week 8.
- Contralateral Unaffected Skin: Change in bacterial load in a given sample using log10 (bacterial count/ sample) units at baseline prior to initiation of phototherapy and at week 8 after the initiation of phototherapy.
  Comparison between contralateral unaffected skin at baseline vs contralateral unaffected skin week 8.
- Unaffected Back: Change in bacterial load in a given sample using log10 (bacterial count/ sample) units at baseline prior to initiation of phototherapy and at week 8 after the initiation of phototherapy.
  Comparison between unaffected back at baseline vs unaffected back week 8.
Arm/Group | Plaque Center | Plaque Edge | Ipsilateral Perilesional Unaffected Skin | Ipsilateral Distant Unaffected Skin | Contralateral Unaffected Skin | Unaffected Back
Number analyzed (Participants) | 34 | 18 | 31 | 32 | 16 | 33
Log10 [bacterial count/sample] | 0.53 (0.20) | 0.85 (0.41) | -0.05 (0.23) | -0.08 (0.16) | -0.01 (0.20) | -0.01 (0.18)

9. Primary Outcome: Change in Cutaneous Bacterial Load Between Baseline and Week 9.
Description: Bacterial count per sample at baseline prior to initiation of phototherapy vs at week 9 after initiation of phototherapy.
Time Frame: Week 9
Measure: Mean (Standard Error); unit: Log10 [bacterial count/sample]
Groups:
- Plaque Center: Change in bacterial load in a given sample using log10 (bacterial count/ sample) units at baseline prior to initiation of phototherapy and at week 9 after the initiation of phototherapy.
  Comparison between plaque center at baseline vs plaque center at week 9.
- Plaque Edge: Change in bacterial load in a given sample using log10 (bacterial count/ sample) units at baseline prior to initiation of phototherapy and at week 9 after the initiation of phototherapy.
  Comparison between plaque edge at baseline vs plaque edge at week 9.
- Ipsilateral Perilesional Unaffected Skin: Change in bacterial load in a given sample using log10 (bacterial count/ sample) units at baseline prior to initiation of phototherapy and at week 9 after the initiation of phototherapy.
  Comparison between ipsilateral perilesional unaffected skin at baseline vs ipsilateral perilesional unaffected skin at week 9.
- Ipsilateral Distant Unaffected Skin: Change in bacterial load in a given sample using log10 (bacterial count/ sample) units at baseline prior to initiation of phototherapy and at week 9 after the initiation of phototherapy.
  Comparison between ipsilateral distant unaffected skin at baseline vs ipsilateral distant unaffected skin at week 9.
- Contralateral Unaffected Skin: Change in bacterial load in a given sample using log10 (bacterial count/ sample) units at baseline prior to initiation of phototherapy and at week 9 after the initiation of phototherapy.
  Comparison between contralateral unaffected skin at baseline vs contralateral unaffected skin week 9.
- Unaffected Back: Change in bacterial load in a given sample using log10 (bacterial count/ sample) units at baseline prior to initiation of phototherapy and at week 9 after the initiation of phototherapy.
  Comparison between unaffected back at baseline vs unaffected back week 9.
Arm/Group | Plaque Center | Plaque Edge | Ipsilateral Perilesional Unaffected Skin | Ipsilateral Distant Unaffected Skin | Contralateral Unaffected Skin | Unaffected Back
Number analyzed (Participants) | 34 | 18 | 31 | 32 | 16 | 33
Log10 [bacterial count/sample] | 0.68 (0.17) | 0.61 (0.42) | -0.01 (0.17) | -0.01 (0.15) | -0.02 (0.24) | -0.002 (0.18)

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | NB-UVB Phototherapy
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 17/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NB-UVB Phototherapy (N=34)
Erythema (Skin and subcutaneous tissue disorders) | 14
Tenderness (Skin and subcutaneous tissue disorders) | 12
Burn (Skin and subcutaneous tissue disorders) | 3
Pruiritis (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Statistical Analysis Plan (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT02552316/SAP_000.pdf
  • Study Protocol (2015-09-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT02552316/Prot_001.pdf
  • Informed Consent Form (2016-03-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT02552316/ICF_002.pdf